CLINICAL TRIAL: NCT05694377
Title: Effects of the Electroencephalography-based Neurofeedback Training on Cognitive Function in Healthy Young Men
Brief Title: Effects of the EEG-neurofeedback on Cognitive Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Wroclaw University of Health and Sport Sciences (Other)
Responsible Party: Principal Investigator, Jaroslaw Marusiak, Principal Investigator - Director of Kinesiology Department at the University School of Physical Education in Wroclaw, Wroclaw University of Health and Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 01/2019
Record Dates: First submitted 2023-01-06; First posted 2023-01-23 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Cognitive Function; Executive Function
Keywords: neurofeedback; attention index; cognitive function

STUDY DESIGN:
Intervention Model Description: two arms repeated measures control design
Who Masked: Outcomes Assessor
Masking Description: The person analysing the outcomes will be blinded to the subjects allocation to the groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TR group (Experimental): The training group (TR) will undergo 3 weeks of electroencephalography-based neurofeedback (EEG-NFB). EEG-NFB training.
  Interventions: Behavioral: electroencephalography-based neurofeedback (EEG-NFB)
- CO group (No Intervention): Control group (CO) will not undergo 3 weeks of EEG-NFB training.

INTERVENTIONS:
Behavioral: electroencephalography-based neurofeedback (EEG-NFB) — The EEG-NFB training program will involve nine training sessions (three times a week over a 3-week period) each lasting 30 min. EEG-NFB training will be conducted with ProComp Infiniti Encoder and BioGraph Infiniti Software v.5.1.3. The training protocol will be set to decrease the EEG TBR value. For the 12 training sessions, all participants will be subjected the same EEG-NFB protocol at C3 electrode. The EEG-NFB training sessions consists of a 20-s baseline period (i.e., with no feedback), 30-min feedback presentation, and another 20-s baseline period. Subjects will be seated in front of a computer screen and animations will be used as feedback; the animation starts when the subject is sufficiently focused for 20 s. Three 10-min animations (flying duck, roller coaster ride, and moving ball) will be shown to the subject during each EEG-NFB training session. The raw EEG signal, TBR value over time, EEG signal noise, and EEG theta and beta wave amplitudes will be recorded.
  Arms: TR group

SUMMARY:
Executive function play a key role in boosting human behavioural performance. Based on scientific literature, it is still controversial whether electroencephalography-based neurofeedback (EEG-NFB) represents an effective technique for enhancing healthy adults' executive function. This study evaluates generalized effects of 3-week EEG-NFB training, using self-regulation of the theta to beta wave ratio (TBR), on executive function in healthy adults. The subjects are an uniform group of healthy young right-handed males divided into two equal groups. The trained group (TR) performs 3-week EEG-NFB training (three sessions per week) focused on a cognitive self-regulation of TBR (to achieve the lower TBR values as beneficial cognitive effect), while the control group (CO) does not participate in the EEG-NFB training. Cognitive function are rated before and after 3-week EEG-NFB training by psychological tests: Trail Making Test (TMT, parts A and B) and the Stroop Test (ST, parts I and II). This project is important for the future development of effective EEG-NFB protocols to be used by healthy people to improve their behavioural performance.

DETAILED DESCRIPTION:
2. MATERIALS AND METHODS

2.1. Subjects A total of 50 healthy male students will be randomly assigned to one of two groups of 25 subjects each using a computerized randomization method. The trained group will undergo 3 weeks of EEG-NFB training, whereas the control group will not undergo training. Inclusion criteria for study participation will be lack of any neurological disorders and motor or cognitive deficits, lack of neurological incident in the past, age between 20 to 25 years, male sex, and right-handedness (this inclusion criteria will be to avoid an influence of lateralization and gender on psychological tests outcomes). The study was approved by the ethic committee of the University School of Physical Education in Wroclaw and will be carried out in accordance with the principles outlined in the Declaration of Helsinki.

2.2. Experimental procedure TR and CO groups will be each tested twice in the same time periods, i.e., before 3 weeks period of EEG-NFB training (PRE) and after the training period (POST). During the PRE and POST experimental sessions, all subjects will undergo psychological testing to evaluate executive function. PRE testing in the both groups will be performed 1 to 4 days before the first day of EEG-NFB training period, whereas POST testing will be performed 1 to 4 days after the last day of EEG-NFB training period to ensure that the measurements will be not due to the effects of the last single training session in the TR group.

2.3. Psychological assessment All subjects will undergo cognitive testing (TMT and ST), which will be performed by an experienced researcher. There will be two parts to the TMT: TMT-A, in which a subject connects numbers in sequential order; and TMT-B, in which the subject alternates between numbers and letters (1, A, 2, B, etc.). The former is used to examine cognitive processing speed, while the latter assesses executive function. The ST also consists of two parts: ST-I, in which a subject reads a list of 40 words, which are names of colours printed in the colour itself; and ST-II, where colour names are printed in an incongruent colour and the subject is required to ignore the word and correctly name the ink colour. The former is used as a measure of processing speed and the latter to test selective attention and inhibition. The subjects will be provided with instructions prior to starting the TMT and ST. In both ST tests parts subjects will have the same instruction as "name the colour of ink", and will not be informed in ST-I that all name/ink are matched. All tests (both parts of TMT and ST) will be preceded by preparatory/training trials, a similar but shorter version of main tests. Before starting each test, subjects will be instructed to concentrate and to make use their maximal attention skills during testing session. In both tests (TMT and ST), the time taken to complete the test will be used as the performance measure, with a shorter time reflecting a better performance. The tests will be administered in a quiet room with only one and always the same investigator present.

2.4. EEG-NFB training procedure The EEG-NFB training program will involve nine training sessions (three times a week over a 3-week period) each lasting 30 min. EEG-NFB training will be conducted with ProComp Infiniti Encoder and BioGraph Infiniti Software v.5.1.3. The training protocol will be set to decrease the EEG TBR value. For the 12 training sessions, all participants will be subjected the same EEG-NFB protocol at C3 (according to the 10-20 system), which is related to Brodmann area 4. This location is selected because the TMT and ST used to quantify the EEG-NFB effect are also related to activity in this brain region. The EEG-NFB training sessions consists of a 20-s baseline period (i.e., with no feedback), 30-min feedback presentation, and another 20-s baseline period. Subjects will be seated in front of a computer screen and animations will be used as feedback; the animation starts when the subject is sufficiently focused for 20 s. Three 10-min animations (flying duck, roller coaster ride, and moving ball) will be shown to the subject during each EEG-NFB training session. The raw EEG signal, TBR value over time, EEG signal noise, and EEG theta and beta wave amplitudes will be recorded.

TBR values will be recorded and calculated for each training session for the TR group and will be compared between the beginning of the first and beginning of the last EEG-NFB training sessions, to determine whether the 3-week training lead to decrease of the TBR value.

2.5. Statistical analysis The Shapiro-Wilk test will be used to estimate the distribution of psychological parameters. The Wilcoxon signed-rank test or Student's t-test will be used to assess the statistical significance of differences for paired sample comparisons (i.e., between PRE and POST testing sessions). The Mann-Whitney test or Student's t-test will be used for unpaired sample comparisons (i.e., between TR and CO groups). Magnitude/importance of differences will be calculated using the Cohen effect size d value for results of the psychological tests; a value of 0 indicates no effect, whereas values > 0.2, >0.6, and > 0.8 indicates small, moderate, and large effects, respectively. P value ≤ 0.05 will be taken as statistically significant for all analyses. All statistical analyses will be performed using SPSS Statistics 22.0 software (IBM, Armonk, NY, USA).

ELIGIBILITY:
Inclusion Criteria:

* lack of any neurological disorders including motor or cognitive deficits
* right-handedness

Exclusion Criteria:

* diagnosed neurological disorders including motor or cognitive deficits
* left-handedness

Ages: 20 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — participant eligibility is based on self-representation
Enrollment: 60 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
TMT-A | 1 week prior EEG-NFB training program
  trail making test, part A is a psychological measure of cognitive processing speed, measured as performance time (the shorter the time the better performance), expressed in [s].
TMT-A | up to 1 week post EEG-NFB training program
  trail making test, part A is a psychological measure of cognitive processing speed, measured as performance time (the shorter the time the better performance), expressed in [s].
TMT-B | 1 week prior EEG-NFB training program
  trail making test, part B is a psychological measure of executive function, measured as performance time (the shorter the time the better performance), expressed in [s].
TMT-B | up to 1 week post EEG-NFB training program
  trail making test, part B is a psychological measure of executive function, measured as performance time (the shorter the time the better performance), expressed in [s].
ST-I | 1 week prior EEG-NFB training program
  Stroop Test, part I is used as a psychological measure of processing speed, measured as performance time (the shorter the time the better performance), expressed in [s].
ST-I | up to 1 week post EEG-NFB training program
  Stroop Test, part I is used as a psychological measure of processing speed, measured as performance time (the shorter the time the better performance), expressed in [s].
ST-II | 1 week prior EEG-NFB training program
  Stroop Test, part II is used as a psychological measure of selective attention and inhibition, measured as performance time (the shorter the time the better performance), expressed in [s].
ST-II | up to 1 week post EEG-NFB training program
  Stroop Test, part II is used as a psychological measure of selective attention and inhibition, measured as performance time (the shorter the time the better performance), expressed in [s].

CONTACTS AND LOCATIONS:
Overall Officials: Malgorzata Slowinska-Lisowska, Study Director — Wroclaw University of Health and Sport Sciences
Locations (1):
- University School of Physical Education in Wroclaw, Wroclaw, Lower Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
Only anonymized data will be shared with other researchers based on their request to principal investigator.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be available from January the the 1'st of 2024.
Access Criteria: Data will be shared with other researchers based on their request to principal investigator.
URL: http://awf.wroc.pl